CLINICAL TRIAL: NCT00010816
Title: Herbal Treatment of Hepatitis C in Methadone Maintained Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: P50AT000009-02P3 (NIH); P50AT000009-02 (NIH); P50AT000009-03 (NIH); NCT00009464 (obsolete NCT alias)
Record Dates: First submitted 2001-02-02; First posted 2001-02-05 (Estimated); Last update posted 2006-08-18 (Estimated); Status verified 2006-08

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C

INTERVENTIONS:
Drug: Herbal remedies

SUMMARY:
Hepatitis C (HCV) is a chronic viral illness leading to progressive liver damage that has emerged as a major public health issue in the United States. While HCV affects all population groups, individuals with a history of intravenous drug use form the largest known risk group. Between 90 and 100 percent of long term intravenous drug use will eventually test positive for HCV, and there is substantial risk that even short term experimentation will result in infection. Studies suggest that HCV will be the major cause of cirrhosis and liver cancer in the next century. Currently, approved therapy includes recombinant interferons, which lead to sustained remission in a minority of patients. However, patients abusing other substances, including alcohol, are not eligible for interferon therapy. The need for investigation into other potential therapies is clear. Current practice patterns in the Far East include the use of traditional herbal remedies for symptomatic chronic viral hepatitis. This study is intended to examine the effect of commonly used herbal remedies for the treatment of symptomatic HCV.

ELIGIBILITY:
Inclusion Criteria:

* English speaking/reading
* Serum positive for HCV virus by PCR
* Elevated alanine transferase (ALT) within 6 months of the Entry Visit, unattributable to causes other than HCV
* Liver biopsy within 2 years of entry confirming that the histological diagnosis is consistent with chronic HCV
* Laboratory parameters available at the Entry Visit including CBC, differential, and platelet count.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1998-09; Study Completion 2003-06

CONTACTS AND LOCATIONS:
Overall Officials: Jeff Albrecht, MD, Principal Investigator — Hennepin County Medical Center, Minneapolis
Locations (1):
- Hennepin County Medical Center, Minneapolis, Minnesota, United States